CLINICAL TRIAL: NCT02884232
Title: Application of Guidelines for Medico-professional Supervision of Workers Exposed to Carcinogenic Action of Wood Dust: CERBois Cohort. Feasibility Evaluation
Brief Title: Application of Guidelines for Medico-professional Supervision of Workers Exposed to Carcinogenic Action of Wood Dust: CERBois Cohort
Acronym: CERBois
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/INCA/CERBOIS/PARIS-HERIN
Record Dates: First submitted 2016-08-23; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Exposition to Wood Dust

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Workers exposed to wood dust
  Interventions: Procedure: Nasofibroscopy

INTERVENTIONS:
Procedure: Nasofibroscopy

SUMMARY:
The purpose is to evaluate feasibility of medical supervision of professionally active asymptomatic wood workers with questionnaires and nasofibroscopy.

Secondary purposes are:

* Feasibility evaluation of identification of former and actual professional expositions to wood dust and to various naso-sinusal carcinogenics in case of co-expositions (formaldehyde, chrome, nickel, leather)
* Description of abnormal symptoms identified by occupational doctor and needing an otorhinolaryngology test
* Description of results and examinations induced by nasofibroscopy in symptomatic or asymptomatic individuals: counting of naso-sinusal adenocarcinoma cases
* Evaluation of participation of workers retiring in 2 years after inclusion to medical supervision program
* Evaluation of information flow among different players
* Assessment of costs induced by this targeted screening: direct medical costs (screened pathologies, induced additional examinations…) and indirect costs for company (duration of worker absence for transfer, medical and additional examinations).

ELIGIBILITY:
Inclusion Criteria:

* Employee or craftsman
* Actual or former professional exposition to wood dust
* Onset of exposition to wood dust back to more than 30 years (latency >30 years)
* Cumulated exposition to wood dust longer than 12 months
* Exposition to wood dust during machining tasks (sawing, milling, planing, drilling, bridging) or all documented activities exposing to wood dust concentration > 1 mg/m3 for 8 hours
* Worker followed by occupational doctor of participant occupational health departments
* Worker accepting medico-professional supervision recommended by guidelines
* Affiliation to social security

Exclusion Criteria:

* Difficulty with comprehension of wood auto-questionnaire

Min Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population under analysis consists of all workers seen in occupational health consultation and exposed to wood dust at least for cumulated 12 months and with first exposition back to more than 30 years
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Participation to medical supervision program of professionally active asymptomatic workers | Day 0
Participation to medical supervision program of professionally active asymptomatic workers | 3 months
Participation to medical supervision program of professionally active asymptomatic workers | 24 months
Participation to medical supervision program of professionally active asymptomatic workers | 27 months

SECONDARY OUTCOMES:
Former and actual professional expositions to wood dust and to various naso-sinusal carcinogenics | Day 0
Presence of abnormal symptoms assessed by doctor, needing an otorhinolaryngology test | Day 0
Presence of abnormal symptoms assessed by doctor, needing an otorhinolaryngology test | 24 months
Counting of diagnoses of naso-sinusal adenocarcinoma in symptomatic and asymptomatic workers after nasofibroscopy | 3 months
Counting of diagnoses of naso-sinusal adenocarcinoma in symptomatic and asymptomatic workers after nasofibroscopy | 27 months
Participation to medical supervision program of workers retiring in 2 years after inclusion | Day 0
Evaluation of information flow among different players | 3 months
Evaluation of information flow among different players | 27 months
Medical costs Induced by screening | 3 months
Medical costs Induced by screening | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PARIS, Pr, Principal Investigator — Centre de Consultations de Pathologies Professionnelles - Hôpitaux de Brabois - CHU de Nancy - France
Locations (6):
- France (6):
  - AHI 33, Bordeaux
  - Pôle Santé Travail, Lille
  - Gnmst-Btp, Paris
  - Ville de Paris, Paris
  - ACMS, Suresnes
  - Centres de Consultations de Pathologies Professionnelles, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No